CLINICAL TRIAL: NCT04411017
Title: Protocol for Optimizing Colonoscopy Preparation in Patients With Inflammatory Bowel Disease
Acronym: EII_Prep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, María Dolores Martín Arranz, PhD, Principal Investigator, Hospital Universitario La Paz
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EII_Prep
Record Dates: First submitted 2019-07-24; First posted 2020-06-01 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2020-05

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Colonoscopy; Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1L PEG (Active Comparator)
  Interventions: Procedure: Endoscopy
- 2L PEG (Active Comparator)
  Interventions: Procedure: Endoscopy
- 2L sodium picosulfate (Active Comparator)
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Colonoscopy

SUMMARY:
Clinical trial evaluating efficacy of bowel cleansing solutions in patients with Inflammatory Bowel Disease.

DETAILED DESCRIPTION:
Simple blind, randomized study evaluating efficacy of 1LPEG vs 2L PEG vs 2L sodium picosulfate in bowel cleansing of patients diagnosed of Inflammatory Bowel Disease undergoing diagnostic or follow-up routine colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18y and 90y
* Patients with a diagnosis of IBD undergoing follow-up or screening colonoscopy

Exclusion Criteria:

* Patients <18y or >90y
* Pregnant Women
* Patients with a past history of inadequate bowel cleansing in a colonoscopy performed in the previous 12 months prior to initiation of study
* Patients with a history of bowel resection
* Patients undergoing therapeutic colonoscopy
* Patients unable to understand study protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Bowel cleansing | 1 year
  Boston Bowel Preparation Score (BBPS), a 10-point scale assessing bowel preparation after all cleansing maneuvers are completed by the endoscopist. Each region of the colon receives a "segment score" from 0 to 3 and these segment scores are summed for a total BBPS score ranging from 0 to 9. Therefore, the maximum BBPS score for a perfectly clean colon without any residual liquid is 9 and the minimum BBPS score for an unprepared colon is 0.

SECONDARY OUTCOMES:
Treatment related adverse events | 1 year
  Number of Participants with symptomatology related to intervention in each arm of the study
Preparation Tolerability: total volume of solution finally taken by the patient | 1 year
  Evaluation of total volume of solution finally taken by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dolores Martin Arranz, PhD, Principal Investigator — Hospital Universitario La Paz. IdiPaz. Universidad Autónoma de Madrid.
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrd, Spain

IPD SHARING:
Plan to Share IPD: No